CLINICAL TRIAL: NCT04306848
Title: Temporary Use of a Continuous Glucose Monitoring System as an Adjunct to Lifestyle Medicine Education for People With Type 2 Diabetes: a Feasibility Study.
Brief Title: Temporary Use of a Continuous Glucose Monitoring System as an Adjunct to Lifestyle Medicine Education
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Software company providing devices never responded. I believe they closed.
Sponsor: Ohio University (Other)
Collaborators: Memorial Health System (Other)
Responsible Party: Principal Investigator, David Drozek, Associate Professor, Ohio University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBD-2
Record Dates: First submitted 2020-03-11; First posted 2020-03-13 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Blood Glucose Profile
Keywords: continuous glucose monitoring, lifestyle medicine

STUDY DESIGN:
Intervention Model Description: Pilot / feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Pilot (Experimental): Eligible subjects who have consented to the study, and have had the baseline data gathered as part of their participation in the Lifestyle Medicine Clinic, an intensive therapeutic lifestyle medicine program, will be given a CGMs device and supplies, and instructed in how to utilize these. They will set up the app on their smart phone to provide them with feedback on their glucose level to correlate with their lifestyle activities.
  Interventions: Device: Temporary Continuous Glucose Monitoring System

INTERVENTIONS:
Device: Temporary Continuous Glucose Monitoring System — This is a feasibility study evaluating the potential to utilize a continuous glucose monitoring system (CGMs) on a temporary basis, during participation in an intensive therapeutic lifestyle medicine program, to help improve the compliance with healthy lifestyle changes for people with Type 2 diabetes (T2DM) and prediabetes (PD).
  Other Names: Intensive therapeutic lifestyle medicine

SUMMARY:
This is a feasibility study evaluating the potential to utilize a continuous glucose monitoring system (CGMs) on a temporary basis, during participation in a lifestyle medicine program, to help improve the compliance with healthy lifestyle changes for people with Type 2 diabetes (T2DM) and prediabetes (PD).

DETAILED DESCRIPTION:
Glucose peaks after eating are an indication of the level of insulin resistance and the severity of disease in patients with T2DM. Many lifestyle factors affect the glucose elevation, including the glycemic index of food, timing of eating, physical activity, stress and sleep.

In practice, a glycemic profile, consisting of multiple glucose measurements before and after meals throughout the day, has sometimes been helpful in educating patients concerning the effects of their eating habits on blood sugar levels.

Would temporary use (8-10 weeks) of a continuous glucose monitoring system (CGMs) be a useful adjunct during lifestyle education in patients with T2DM or PD?

The purpose of this feasibility study is to evaluate the effectiveness of a CGMs on a small sample of patients while they are enrolled in a lifestyle medicine class, to:

* identify any logistical issue involved
* verify that useful data can be obtained for analysis
* inform development of a larger controlled study

Eligible subjects who have consented to the study, and have had the baseline data gathered as part of their participation in the Lifestyle Medicine Clinic, will be given a CGMs device and supplies, and instructed in how to utilize these. They will set up the app on their smart phone to provide them with feedback on their glucose level to correlate with their lifestyle activities.

The FDA approved CGMs utilizes a small filament-like probe that is entered into the skin and measures sugar levels of the interstitial fluid of the subcutaneous tissue. This correlates with blood glucose levels.

Daily, the subjects will enter data into their smart phone app, which will include:

* time of arising in the morning, and perceived quality of sleep
* time and description of food and beverages consumed
* time and description of physical activity
* time and description of stress management activities
* time and duration of naps
* bedtime

Once daily, the subject will complete a reflection entry in a diary on their glucose levels over the last 24 hours in relation to their logged lifestyle activities.

At the completion of the 8 sessions of The Lifestyle Medicine Clinic, participants will complete a survey asking open ended question concerning the use of the CGMs.

ELIGIBILITY:
Inclusion criteria:

* be able to read and write English.
* be enrolled in The Lifestyle Medicine Clinic, taught by Dr. Drozek
* be diagnosed with type 2 diabetes (T2DM) or prediabetes (PDM)
* be at least 18 years of age
* be comfortable wearing a sensor continuously for up to 10 weeks
* have a smart phone and be comfortable utilizing apps
* be able and willing to daily enter data concerning food consumed, exercise, stress management activities and sleep.
* be willing to complete a daily reflection on the relationship of their blood sugar to lifestyle activities.
* be willing to complete a survey at the completion of the project about their perceptions of utilizing continuous glucose monitoring (CGM)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Blood glucose profile | 12 weeks
  The blood glucose profile will be evaluated for out of range values

SECONDARY OUTCOMES:
participant survey | 12 weeks
  1. Specifically concerning the Diabits software:
     1. What did you like about Diabits?
     2. What didn't you like about Diabits?
     3. Do you think Diabits has improved your blood sugar management?
  2. Did you complete the data entry most of the time? If not, please explain, and make suggestions on how the experience could be improved.
  3. Did you have any difficulty managing the sensor or device? If so, please explain, and make suggestions on how the experience could be improved.
  4. Overall, did you feel that the continuous glucose monitoring system was helpful? Please explain your answer. How was it helpful or unhelpful?
  5. What else should we know or would you like to tell us?

CONTACTS AND LOCATIONS:
Locations (1):
- Marietta Memorial Hospital, Marietta, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data will be posted after completion of the study.